CLINICAL TRIAL: NCT02338479
Title: Natural History and Biology of Long-Term Late Effects Following Hematopoietic Cell Transplant for Childhood Hematologic Malignancies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Pediatric Blood and Marrow Transplant Consortium (Other); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: 13-TLEC
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphoblastic Leukemia/Lymphoma; Myelodysplasia; Acute Myelogenous Leukemia; Juvenile Myelomonocytic Leukemia; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective non-therapeutic study, assessing the long-term toxicity of pediatric HCT for hematologic malignancies. This study is a collaboration between the Pediatric Blood and Marrow Transplant Consortium (PBMTC), the Center for International Blood and Marrow Transplant Research (CIBMTR), the National Marrow Transplant Program (NMDP) and the Resource for Clinical Investigation in Blood and Marrow Transplantation (RCI-BMT) of the CIBMTR. The study will enroll pediatric patients who undergo myeloablative HCT for hematologic malignancies at PBMTC sites.

DETAILED DESCRIPTION:
This is a prospective non-therapeutic study, assessing the long-term toxicity of pediatric HCT for hematologic malignancies. This study is a collaboration between the Pediatric Blood and Marrow Transplant Consortium (PBMTC), the Center for International Blood and Marrow Transplant Research (CIBMTR), the National Marrow Transplant Program (NMDP) and the Resource for Clinical Investigation in Blood and Marrow Transplantation (RCI-BMT) of the CIBMTR. The study will enroll pediatric patients who undergo myeloablative HCT for hematologic malignancies at PBMTC sites.

The study examines the hypothesis that survivors of pediatric HCT are at risk for late organ toxicity and they will have identifiable biomarkers present within the first two years following HCT which will be predictive for late adverse outcomes allowing for early identification of patients at risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 22 years at admission for HCT
2. Planned allogeneic HCT from any donor and stem cell source. There are no study-specific criteria for HLA-matching
3. Disease and disease status criteria

   1. Acute lymphoblastic leukemia/lymphoma in complete morphologic remission defined as a M1 marrow (<5% blasts) with no evidence of active extramedullary disease within 30 days of the start of the conditioning regimen; OR
   2. Myelodysplasia (regardless of subtype) with less than 10% marrow blasts within 30 days of the start of the conditioning regimen; OR
   3. Acute myelogenous leukemia in complete morphologic remission defined as an M1 marrow (<5% blasts) with no evidence of extramedullary disease within 30 days of the start of the conditioning regimen; OR
   4. Juvenile myelomonocytic leukemia; OR
   5. Chronic myelogenous leukemia excluding refractory blast crisis.
4. Planned myeloablative conditioning regimen, defined as a regimen including one of the following as a backbone agent:

   1. Busulfan ≥ 12.8 mg/kg total dose (IV or PO). PK-based dosing allowed, if the intent is total overall dose ≥ 12.8 mg/kg; OR
   2. Total Body Irradiation ≥ 1200 cGy fractionated; OR
   3. Treosulfan ≥ 30 g/m2 total dose IV
5. Enrollment in the following NMDP research protocols:

   1. Protocol for a Research Database for Hematopoietic Cell Transplantation, Other Cellular Therapies and Marrow Toxicity Injuries
   2. Protocol for a Research Sample Repository for Allogeneic Hematopoietic Stem Cell Transplantation and Marrow Toxic Injuries
6. Written informed consent document signed by patient if the age is greater than or equal to 18 years and the patient is developmentally able to provide consent. The informed consent document is to be signed by the parent or legal guardian if the patient's age is less than 18 years or if the patient is older than 18 years, but developmentally unable to provide consent. Assent will be obtained according to the guidelines of the patient's transplant institution.

Exclusion Criteria:

1. Prior allogeneic or autologous HCT
2. Patients with renal disease prior to the start of HCT conditioning requiring the use of dialysis at the time of enrollment and/or GFR < 60 mL/min/1.73 m2
3. Patients with osteopenia or osteoporosis treated with a bisphosphonate medication at any time prior to enrollment
4. Patients with preexisting diabetes or hyperglycemia treated with insulin or oral hypoglycemic medication at the time of enrollment
5. Patients with uncontrolled viral, bacterial, fungal or protozoal infection at the time of study enrollment
6. Karnofsky performance score or Lansky Play-Performance Scale Score <60 at the time of study enrollment
7. Known inherited or constitutional predisposition to cancer including, but not limited to Down Syndrome, Li-Fraumeni syndrome, Fanconi Anemia, and patients with BRCA1 and BRCA2 mutations

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll is a nonrandomized prospective cohort undergoing HCT for treatment of childhood leukemia and myelodysplasia.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To report the incidence of chronic kidney disease (CKD), metabolic syndrome, and osteopenia | Baseline to 1 and 2 years following allogeneic HCT for hematologic malignancy

SECONDARY OUTCOMES:
To identify prognostic risk factors for the development and progression of post-HCT CKD, metabolic syndrome, and osteopenia | Baseline to 1 and 2 years following HCT
To investigate potential associations of systemic hypertension as measured with intermittent blood pressure assessment with proteinuria, acute kidney injury, and CKD | Baseline to 100 days, and at 1 and 2 years following HCT
To compare the results of GFR estimating equations based on serum cystatin C levels or serum creatinine to GFR measured by nuclear medicine GFR and/or 24-hour creatinine clearance | Baseline to 180 days, and at 1 and 2 years following HCT
To explore potential association of the protein biomarker elafin in the urine at with the development of CKD | Baseline to 180 days, and at 1 and 2 years following HCT
To report levels of fasting triglycerides, low-density lipoprotein, high-density lipoprotein, insulin, and glucose levels | Baseline to 100 days, and at 1 and 2 years following HCT
To assess change in body composition including bone mineral density, body mass index, percent fat mass and lean body mass as measured by dual-energy absorptiometry | Baseline to 1 and 2 years following HCT
To assess the presence of osteopenia prior to HCT and at 1-year and 2-years following HCT by x-ray in patients unable to undergo DXA without sedation | Baseline to 1 and 2 years following HCT
To report levels of markers of bone turnover including serum osteocalcin, bone specific alkaline phosphatase, and urine N-telopeptide | Baseline to 30 days, 100 days, and at 1 and 2 years following HCT
To develop a repository for plasma to be used in future investigation of HCT-associated late effects | Baseline, 30 days, 100 days, and at 1 and 2 years following HCT

CONTACTS AND LOCATIONS:
Overall Officials: Christine Duncan, MD, Study Chair — Dana-Farber Cancer Institute; K. Scott Baker, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (32):
- United States (32):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCLA Center for Health Sciences, Los Angeles, California
  - Children's Hospital & Research Center - Oakland, Oakland, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Hospital/Riley Hospital for Children, Indianapolis, Indiana
  - Dana Farber Cancer Institute - Pediatrics, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - The Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center - Pediatrics, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University - Doernbecher Children's Hospital, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin